CLINICAL TRIAL: NCT07254624
Title: Glucosidase Inhibitors and Glucose Metabolism
Brief Title: Pilot Assessment of Continuous Glucose Monitor for Post-meal Glucose Responses to Herbs and Spices.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: McCormick Science Institute (Industry)
Responsible Party: Principal Investigator, Daniel L. Smith, Jr., Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB-300015105; McCormick Science Institute (Other Grant/Funding Number: McCormick Science Institute)
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Post-prandial Glucose Response
Keywords: post-meal glucose response
MeSH Terms: interventions — Spices

STUDY DESIGN:
Intervention Model Description: Participants will serve as their own controls in this study. They will be randomized to the order they receive the prepared entrees. Post-prandial glucose responses will be compared across the three entree types.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Potato entree with no herbs or spices (Sham Comparator): consumption of a standardized potato entree, matched for macronutrient, calorie and preparation method across arms
  Interventions: Other: Potato entree
- Potato entree with herbs or spices (Experimental): consumption of a standardized potato entree including a mix of five herbs and spices at a fixed amount, matched for macronutrient, calorie and preparation method across arms
  Interventions: Other: Mix of five herbs and spices; Other: Potato entree
- Potato entree with no herbs or spices, with herbs and spices mix at a subsequent meal (Sham Comparator): consumption of a standardized potato entree, matched for macronutrient, calorie and preparation method across arms - with a provision including a mix of five herbs and spices at a fixed amount to be consumed at a subsequent meal within the same day (>2 hours following the potato entree consumption)
  Interventions: Other: Mix of five herbs and spices; Other: Potato entree

INTERVENTIONS:
Other: Mix of five herbs and spices — Herb and spice blend of dried oregano, basil, rosemary, garlic powder and onion powder
  Arms: Potato entree with herbs or spices; Potato entree with no herbs or spices, with herbs and spices mix at a subsequent meal
Other: Potato entree — A potato entree with a fixed macronutrient and calorie content, and standardized preparation method to evoke a post-prandial glucose response

SUMMARY:
The purpose of this study is to determine whether continuous glucose monitoring is sensitive to quantifying the glucose response related to consumption of a starchy vegetable (potato) in combination with or separate from consumption of herbs and spices at the same meal.

DETAILED DESCRIPTION:
This is a pilot study which will enroll a maximum of 10 participants. There will be 3 different food entree preparations that participants will consume (1 entree per day within the 10 day period). The order in which participants eat the different entrees will be randomized. The 3 different food entree preparations are as follows: 1) prepared potato entree with no herbs and spices, 2) prepared potato entree paired with herbs and spices, 3) prepared potato entree with herbs and spices consumed at a subsequent meal.

Following enrollment, participants will be randomized to the order of entree preparation types and provided all of the entrees with the instructions for food preparation and order of consumption noted when they arrive at the scheduled study visit. The entrees will be standardized for caloric content, composition, and preparation method. Post-consumption glucose responses will be recorded by continuous glucose monitors, which will be provided to participants at the first study visit.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI): 20-35
* no dietary restriction or food allergies to study items
* weight stable
* access to a smart phone
* willingness to wear a continuous glucose monitor for the duration of the study (at minimum 10 days)

Exclusion Criteria:

* pregnancy or anticipating pregnancy or lactation
* food allergy to study items
* diagnosed diabetes (type 1 or 2) or taking diabetes medications
* history of bariatric surgery
* consumed >1 serving of potatoes daily before enrollment
* 5% weight loss or gain within the past 6 months
* medical conditions or medication that would prevent the ability to comply with the treatment assignment and/or affect blood glucose or energy balance
* condition which would prevent the ability to wear a continuous glucose monitor on the upper arm for the study duration

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Post-prandial glucose response | 0, 1, and 2 hours post-meal, as well as 24 hour continuous
  Glucose response will be measured using continuous glucose monitors. These devices will capture changes in glucose response from the start of the meal to about 2 hours postprandial.

SECONDARY OUTCOMES:
Acceptance assessment | 0-10 days
  Feedback surveys to assess meal items likeability/acceptability, adherence and feasibility ('1-5' point scale, with '3' being 'neutral' and '5' indicating the participants 'strongly agree' with regarding the likeability and acceptability of the food item) in preparation for a full trial.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data will be shared or made publicly available for any publication of findings.
Time Frame: Following publication of results
Access Criteria: Public repository